CLINICAL TRIAL: NCT01029041
Title: Stretching and Strengthening Exercise in Treatment of Fibromyalgia Patients: a Randomized Clinical Trial
Brief Title: Stretching and Strengthening Exercise in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ana Assumpção Berssaneti, Medicine School of University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cappesq 0337/07
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-12

CONDITIONS: Fibromyalgia Syndrome
Keywords: fibromyalgia, exercise, strength, stretch
MeSH Terms: conditions — Fibromyalgia; Motor Activity | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Strengthening exercise (Experimental): This group does global strengthening exercise
  Interventions: Other: Strengthening Exercises
- Stretching exercise (Experimental): This group does global stretching exercise
  Interventions: Other: Stretching exercises
- Control (No Intervention): This group does nor do any kind of exercise during the study

INTERVENTIONS:
Other: Strengthening Exercises — Exercises that aim the improvement of muscular strength of arms and legs
  Other Names: strengh exercise
  Arms: Strengthening exercise
Other: Stretching exercises — Exercises that aim the improvement of muscular flexibility of arms, legs and spine
  Other Names: flexibility exercise
  Arms: Stretching exercise

SUMMARY:
Fibromyalgia is a rheumatologic syndrome characterized by widespread chronic pain, tender points and other symptoms as fatigue, sleep disturbances, anxiety and depression. Therapeutic exercises are described as an important form to management of symptoms. This study aims to assess strengthening and stretching exercise efficacy in symptoms and quality of life of Fibromyalgia patients. The study is done at General Clinical Hospital of Medicine Scholl of University of Sao Paulo. 63 subjects undergo the study and they are divided into three groups: 1 strengthening exercise, 2 stretching exercise and 3 control group. Patients are evaluated by following instruments: Fibromyalgia Impact Questionnaire, Medical Outcomes Study 36-item Short-Form Health Survey (SF-36), Stanford Health Assessment Questionnaire, dolorimetry at tender points by a Fischer dolorimeter, finger-to-tip floor test for muscular flexibility, dynamometer EMG System do Brasil for strength test of extension and flexion of knees and elbows, time to get up and go test, functional reach test, sit-to-stand test. Subjects of 1 strengthening exercise group undergo a global strengthening program and 2 stretching exercise group undergo a global stretching program. All programs have 12 weeks of duration and physical therapy is twice a week. The control group does not do any intervention during 12 weeks and after the second evaluation they enter the common program of physical therapy. Data are being analyzed by descriptive and interferential statistics procedures.

DETAILED DESCRIPTION:
In this study, were included subjects with fibromyalgia diagnosis aged between 30 and 55 years old. We aimed to assess the effect of a physical therapy program on impact of fibromyalgia syndrome and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Fibromyalgia diagnosis according to American Rheumatology Criteria
* Aged between 30 and 55 years old

Exclusion Criteria:

* Severe rheumatologic syndromes
* neurologic syndromes

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2007-08; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Fibromyalgia Impact Questionnaire | before and after treatment

SECONDARY OUTCOMES:
Medical Outcomes Study 36-item Short-Form Health Survey (SF-36), Stanford Health Assessment Questionnaire | before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Amélia P Marques, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Medicine School of University of Sao Paulo, São Paulo, São Paulo, Brazil